CLINICAL TRIAL: NCT00516698
Title: Changes in Breast Density and Plasma Hormone Levels After One Year of Aromatase Inhibitor Therapy
Brief Title: Changes in Breast Density and Blood Hormone Levels in Postmenopausal Women Receiving Anastrozole or Exemestane for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-N063I; NCI-2012-02719 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000560200 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis; Chromatography, High Pressure Liquid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients undergo blood sample collection at baseline and at 1 year after initiation of aromatase inhibitor therapy (anastrozole or exemestane). Samples are analyzed for estrogen and testosterone levels and additional hormone levels and growth factors that have been previously linked with breast density and that could be altered by aromatase inhibitor use (i.e., sex hormone-binding globulin [SHBG], DHEA, DHEA sulfate, progesterone, prolactin, insulin-like growth factor-1 [IGF-1], and insulin-like growth factor binding protein 3 [IGF BP3]). Samples are also analyzed for anastrozole and exemestane levels by HPLC. Pharmacogenetic studies are also performed. Haplotype-tagged single nucleotide polymorphisms in genes in the aromatase pathway are examined.
  Patients also undergo mammogram at baseline (≤ 6 months prior to study registration) and at 1 year after initiation of aromatase inhibitor therapy.
  Interventions: Genetic: polymorphism analysis; Other: high performance liquid chromatography; Other: laboratory biomarker analysis; Procedure: radiomammography

INTERVENTIONS:
Genetic: polymorphism analysis
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Procedure: radiomammography

SUMMARY:
RATIONALE: Studying changes in breast density and blood hormone levels in women receiving anastrozole or exemestane for breast cancer may help doctors learn more about the long-term effects of treatment and may help the study of breast cancer in the future.

PURPOSE: This clinical trial is studying changes in breast density and blood hormone levels in postmenopausal women receiving anastrozole or exemestane for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the changes in percent breast density (in response to 1 year of aromatase inhibitor therapy) from levels prior to the initiation of treatment.
* To assess the changes in dense area (in response to 1 year of aromatase inhibitor therapy) from levels prior to the initiation of treatment.
* To examine whether changes in percent breast density (in response to 1 year of aromatase inhibitor therapy) from pre-treatment levels correlate with changes in plasma hormone levels (estrone, estrone-sulfate, estradiol, and SHBG) and drug levels (anastrozole or exemestane) over the same time period.
* To examine whether changes in dense area (in response to 1 year of aromatase inhibitor therapy) from pre-treatment mammogram correlate with changes in plasma hormone levels (estrone, estrone-sulfate, estradiol, and SHBG) and drug levels (anastrozole or exemestane) over the same time period.
* To assess whether women with high pre-treatment percent density (upper tertile) experience greater decreases in percent breast density after 1 year of aromatase inhibitor therapy than women with low pre-treatment percent density (lower tertile).
* To assess whether women with high pre-treatment dense area (upper tertile) experience greater decreases in dense area after 1 year of aromatase inhibitor therapy than women with low pre-treatment dense area (lower tertile).
* To examine the associations of haplotype-tagged single nucleotide polymorphisms in genes in the aromatase pathway identified through the Mayo Clinic and Indiana University Pharmacogenomics Research Network Projects, with changes in percent and area density, plasma hormone levels, and drug levels after 1 year of aromatase inhibitor therapy.

OUTLINE: This is a multicenter study.

Patients undergo blood sample collection at baseline and at 1 year after initiation of aromatase inhibitor therapy (anastrozole or exemestane). Samples are analyzed for estrogen and testosterone levels and additional hormone levels and growth factors that have been previously linked with breast density and that could be altered by aromatase inhibitor use (i.e., sex hormone-binding globulin [SHBG], DHEA, DHEA sulfate, progesterone, prolactin, insulin-like growth factor-1 [IGF-1], and insulin-like growth factor binding protein 3 [IGF BP3]). Samples are also analyzed for anastrozole and exemestane levels by HPLC. Pharmacogenetic studies are also performed. Haplotype-tagged single nucleotide polymorphisms in genes in the aromatase pathway are examined.

Patients also undergo mammogram at baseline (≤ 6 months prior to study registration) and at 1 year after initiation of aromatase inhibitor therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Must have histologically confirmed invasive breast cancer, as defined by the following TNM staging criteria:

  * pT1, pT2, or pT3
  * pNx, pN0, pN1, pN2, or pN3*

    * Patients with positive sentinel node biopsies (pN1) must have subsequent axillary dissection to be eligible
    * Patients with negative sentinel node biopsies (pN0) do not require axillary surgery for study eligibility
  * M0, according to the following radiologic studies:

    * Bone scan (required only if alkaline phosphatase is > 2 x institutional upper limit of normal [ULN] and/or there are symptoms of metastatic disease)

      * A confirmatory x-ray or other imaging study, such as CT scan or MRI, is required if the results from the bone scan are questionable
    * Abdominal ultrasound or CT scan of the abdomen (required only if AST/ALT or alkaline phosphatase is > 2 x ULN unless the elevation is in the bone fraction)
    * Chest x-ray NOTE: *Only when the sole basis for this classification is the presence of 10 or more involved axillary nodes
* Completely resected disease

  * Surgical margins must be clear of invasive carcinoma and ductal carcinoma in situ or lobular carcinoma in situ
* Must have one intact, noncancerous breast with no history of previous breast surgery in that breast (other than a breast biopsy)

  * Mammogram of the intact, noncancerous breast required ≤ 6 months prior to study registration (both a craniocaudal [top down] and mediolateral oblique view [side view] must be available)
* Must be registered on this study ≥ 3 weeks but ≤ 3 months after completion of chemotherapy OR primary surgery*

  * Adjuvant chemotherapy and radiation therapy as prescribed by the local institution is allowed provided patient is registered on this study and hormonal treatment is begun as soon as patient has sufficiently recovered from chemotherapy NOTE: *Primary surgery is defined as the last surgical procedure to remove invasive or in situ disease
* Planning to receive anastrozole or exemestane for ≥ 1 year for treatment of breast cancer
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive (defined as a tumor receptor content of > 10 fmol/mg protein OR receptor-positive by immunohistochemistry [ERICA or PgRICA])

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Postmenopausal, defined by one of the following:

  * Age > 60 years
  * Age 45-59 years with spontaneous cessation of menses > 12 months prior to chemotherapy (if no chemotherapy was given, then prior to study registration)
  * Age 45-59 years with cessation of menses for a duration of < 12 months or secondary to hysterectomy AND an FSH level in the postmenopausal range (or ≥ 34.4 IU/L, if institutional range is not available) prior to chemotherapy (if no chemotherapy was given, then prior to study registration)
  * Age 45-59 years with an FSH level in the postmenopausal range according to institutional laboratory standards (or > 34.4 IU/L, if the institutional range is not available) prior to chemotherapy (if no chemotherapy was given, then prior to study registration)
  * Bilateral oophorectomy
* ECOG performance status 0, 1, or 2
* Life expectancy ≥ 5 years

Exclusion criteria:

* History of other (non-breast) malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other curatively treated solid tumors with no evidence of disease for > 5 years
* Any co-existing medical or psychiatric condition that is likely to interfere with study procedures and/or results

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Hormone replacement therapy, oral contraceptives, tamoxifen, raloxifene, other selective estrogen-receptor modulators, or gonadotropin releasing-hormone analogues ≤ 6 months prior to the pre-registration mammogram
* Prior treatment with an aromatase inhibitor (e.g., anastrozole, exemestane, letrozole)
* Planned surgery (other than core needle biopsy) to intact non-cancerous breast (e.g., preventive/prophylactic mastectomy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in percent breast density in response to 1 year of aromatase inhibitor therapy | Up to 12 months
Changes in dense area in response to 1 year of aromatase inhibitor therapy | Up to 12 months
Correlation of changes in percent breast density with changes in plasma hormone levels and drug levels | Up to 12 months
Correlation of changes in dense area with changes in plasma hormone levels and drug levels | Up to 12 months
Comparison of percent breast density in women with high pre-treatment percent density vs women with low pre-treatment percent density | Up to 12 months
Comparison of dense area in women with high pre-treatment dense area vs women with low pre-treatment dense area | Up to 12 months
Associations of haplotype-tagged single nucleotide polymorphisms in genes in the aromatase pathway with changes in percent and area density, plasma hormone levels, and drug levels after 1 year of aromatase inhibitor therapy | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, MD, Study Chair — Mayo Clinic
Locations (180):
- United States (180):
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Southlake Clinic, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming